CLINICAL TRIAL: NCT04458441
Title: Does Warm Skin Disinfection Reduce the Pain Score or Increase the Application Success in Peripheral Central Catheter Application in Premature Babies?
Brief Title: Can Warm Skin Disinfection Reduce the Pain Peripheral Central Catheter Application in Premature Babies?
Acronym: w-pi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Collaborators: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Yavanoglu Atay, principal investigator, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1001
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-07

CONDITIONS: Pain, Acute; Premature
Keywords: premature, pain score, Picc line
MeSH Terms: conditions — Acute Pain; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warm skin desenfection group (Active Comparator): Povidion iodine will be used as a skin cleanser. povidion iodine will be heated sterile to 38 degrees with a ben-mari method and its temperature will be controlled by degrees. When it reaches the appropriate degree, the skin cleaning of the baby will be done sterile.
  Interventions: Other: warm group/cold group
- cold skin desenfection group (No Intervention): Povidion iodine will be used as a skin cleanser. povidion iodine will be used in the skin cleaning of the baby without any heating procedure.

INTERVENTIONS:
Other: warm group/cold group — sequential randomization
  Arms: warm skin desenfection group

SUMMARY:
Peripheral central catheter application, especially in extremely low birth weight premature babies, is an intensive care follow-up procedure. There are many clinical studies in areas such as catheter type, skin disinfection, catheter duration, catheter infection. In our practice, it was observed that premature baby was less uncomfortable, the number of trials decreased, and the change in body temperature was less with the application of hot skin disinfection in our practice. With a prospective randomized study, the investigators wanted to document their observational data scientifically.

DETAILED DESCRIPTION:
Babies under 32 gestation week and 1250 g who are treated at level 3 NICU and need peripheral central catheter will be included in the study. In the preparation of peripheral central catheter application, skin cleaning is performed with povidone iodine in our clinic. The investigators used during the povidione iodine preparation phase after heating the bain-marie method with sterile conditions. The investigators predicted that the premature baby would have less discomfort with warm povidion iodine. To demonstrate this, it was planned to take both video recordings during the application and N-PASS evaluation by an experienced person who does not know the povidone iodine temperature used .In preparation of the catheter except the person who did povidone iodine skin cleansing, nobody knows the heat. The catheters were administered by a single experienced person. The study was designed to be unaware of the povidin iodine application temperature of the person applying the catheter and the N-PASS assessment.

ELIGIBILITY:
Inclusion Criteria: below 32 gestational weeks and / or 1250 grams preterm babies neonates requiring total parenteral nutrition, antibiotic therapy for at least 7 days, -

Exclusion Criteria: major congenital anomalilies refusal to sign consent patient with previously attemped or placed central lines

-

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2022-09-05 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
change feeling of pain and restlessness in premature | every 10 seconds before the 5 minutes and during the procedure
  Evaluation of pain score in the patient during the procedure with n-pass evaluation

SECONDARY OUTCOMES:
protection of body temperature | before 5 min, during procedure
  body temperature monitoring before and during the incubator with skin temperature probe

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Istanbul Umraniye Teaching Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No